CLINICAL TRIAL: NCT00191165
Title: Efficacy and Safety of a High Dosage Compared to the Label Dosage of Humatrope in Early Pubertal Stage Children With Growth Hormone Deficiency
Brief Title: Efficacy and Safety of a High Dosage Compared to the Label Dosage of Somatropin in Early Pubertal Stage Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5202; B9R-IT-GDFU
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-06-08 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Doubled dosage
  Interventions: Drug: Somatropin
- 2 (Active Comparator): In-label dosage
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Doubled dosage with respect to the pre-enrollment (in-label) dosage
  Other Names: LY137998; Humatrope
  Arms: 1
Drug: Somatropin — In-label dosage
  Other Names: LY137998; Humatrope
  Arms: 2

SUMMARY:
Multi-center, randomized, controlled, open-label, phase III study comparing the effects of two different dosages of somatropin treatment (in-label or doubled) after 12 and 24 months of treatment, on height velocity in early pubertal children with growth hormone deficiency (GHD). The study will be conducted in Italy. Approximately 26 subjects will participate in this study, distributed as 13 in the in-label dosage group (group A) and 13 in the doubled dosage group (group B).

ELIGIBILITY:
Inclusion Criteria:

* Height velocity (cm/y) less than 25th percentile at the time of diagnosis.
* diagnosis of GHD
* Replacement therapy at label dosage (from 0.025 to 0.035 mg/kg/day) must be started at least 1 year before the enrolment in this study, but at most 3 years before enrolment
* Bone age less than 12 years for girls and less than 14 years for boys. This assessment should be made by the central reader of bone ages, based on the x-ray taken at Visit 0.
* Informed consent obtained from either both of the subject's parents or legal representative.

Exclusion Criteria:

* Pubertal clinical stage less than 2 and greater than 3 according to Tanner score (for male subjects a volume of testicle greater than 15 mL).
* Any evidence of active malignancy. In case of previous surgical removal of both diencephalic and hypophysial masses, an MRI, performed within six months before enrollment into the study, must exclude the growth of residual tumoral tissue.
* Any known chronic disease such as diabetes mellitus, hepatic disease (defined by elevated liver enzymes 3-fold the upper limit of normal ranges), renal disease with creatinine levels greater than 130 micromol/L, or congestive heart failure.
* Glucocorticoid therapy in supra physiological doses (inhaled corticoids will be accepted if below 3 puffs/day, for no more than 10 days consecutively).
* Current or previous therapy with any therapy that may directly influence growth, including growth hormone releasing hormone, estrogens and anabolic steroids.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2004-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (10):
- Italy (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Novara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Pavia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Torino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Verona

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Somatropin: Somatropin: 0.05 to 0.07 milligram/kilogram/day subcutaneous injection
- Label Dose Somatropin: Somatropin: 0.025 to 0.035 milligram/kilogram/day subcutaneous injection
Period: Overall Study
Arm/Group | High Dose Somatropin | Label Dose Somatropin
Started | 14 | 13
Completed | 12 | 11
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Participant Moved Away | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Somatropin | Label Dose Somatropin | Total
Number analyzed (Participants) | 14 | 13 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 13.5 (1.2) | 13.0 (1.5) | 13.3 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4.0
  Male | 13 | 10 | 23.0
Region of Enrollment [Number; unit: participants]
  Italy | 14 | 13 | 27.0
Race/Ethnicity [Number; unit: participants]
  Caucasian | 14 | 12 | 26.0
  Other | 0 | 1 | 1.0
Baseline Predicted Height [Mean (Standard Deviation); unit: centimeters] — Bone age, chronological age, gender, and height at Visit 0 were used to calculate the Baseline Predicted Height (BLPH) using the method of Bayley and Pinneau.
  Bone age for the BLPH was based on the Greulich-Pyle bone age assessment of the Visit 0 bone age x-ray.
  centimeters | 168 (6.8) | 169 (10.7) | 168 (8.7)
Baseline Predicted Height Standard Deviation Score (SDS) [Mean (Standard Deviation); unit: standard deviation score] — BLPH expressed as a height SDS value (height SDS was derived by subtracting the age-and-gender-matched population 50th percentile height from the patient's height and then dividing this value by the age-and-gender-matched population height standard deviation) using the British standards at age 18 for boys and 16 for girls.
  standard deviation score | -0.9 (0.8) | -0.5 (1.0) | -0.7 (0.9)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter (kg/m2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m2) | 18.9 (3.2) | 19.4 (3.7) | 19.2 (3.4)
Bone Age [Mean (Standard Deviation); unit: years] — Bone age was determined by the Greulich-Pyle method.
  years | 12.4 (0.7) | 12.1 (1.0) | 12.2 (0.8)
Height [Mean (Standard Deviation); unit: centimeters] — Standing measurements were to be made using a standard wall-mounted stadiometer.
  centimeters | 145 (5.1) | 146 (7.8) | 145 (6.5)
Height Standard Deviation Score (SDS) [Mean (Standard Deviation); unit: standard deviation score] — Height SDS was derived by subtracting the age-and-gender-matched population 50th percentile height from the patient's height and then dividing this value by the age-and-gender-matched population height standard deviation (SD).
  standard deviation score | -1.7 (1.0) | -1.1 (1.0) | -1.4 (1.0)
Target Height [Mean (Standard Deviation); unit: centimeters] — Target Height represents the approximate adult height that the patient could be expected to attain, based on the heights of her/his parents. This is a gender-adjusted, average height of the patient's parents' heights calculated in centimeters, modified from the method of Tanner et al.
  centimeters | 168 (5.0) | 168 (7.5) | 168 (6.2)
Target Height Standard Deviation Score (SDS) [Mean (Standard Deviation); unit: standard deviation score] — Target height expressed as height SDS value (see height SDS description for how height SDS value was derived) based on patient's gender, compared to British reference population at age 18 years for males and 16 years for females.
  standard deviation score | -0.9 (0.7) | -0.6 (0.5) | -0.8 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity Standard Deviation Score (SDS) at 12-Month Endpoint
Description: Height velocity (difference between 2 height measurements, divided by years elapsed between measurements) SDS was derived by subtracting age and gender-matched population mean height velocity from patient's height velocity (based on measurements 12 months apart) then dividing this value by age and gender-matched population height velocity SD.
Time Frame: 12-Months
Population: All enrolled participants with baseline and 12-month height measurements.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | High Dose Somatropin | Label Dose Somatropin
Number analyzed (Participants) | 14 | 12
standard deviation score | 1.83 (0.91) | 1.38 (1.41)
Statistical Analysis 1: Comparison: High Dose Somatropin vs Label Dose Somatropin; Test type: Superiority or Other; p = 0.340, ANOVA; Mean Difference (Net) = 0.45, 95% CI [-0.50 to 1.40] — Mean Difference = High Dose - Label Dose

2. Secondary Outcome: Change From Baseline to 12-Month and 24-Month Endpoints in Height Standard Deviation Score (SDS)
Description: This was derived by subtracting the age-and-gender-matched population 50th percentile height from the patient's height and then dividing this value by the age-and-gender-matched population height SD.
Time Frame: Baseline, 12-Months, 24-Months
Population: All enrolled participants with at least one post-baseline height measurement, using last observation available prior to 12-month and 24-month visits respectively, if 12-month or 24-month height was not available.
Measure: Least Squares Mean (Standard Error); unit: standard deviation score
Arm/Group | High Dose Somatropin | Label Dose Somatropin
Number analyzed (Participants) | 14 | 12
standard deviation score
  12-Month Height SDS Change (N=14, N=12) | 0.49 (0.12) | 0.34 (0.13)
  24-Month Height SDS Change (N=13, N=11) | 0.88 (0.17) | 0.40 (0.18)
Statistical Analysis 1: Comparison: High Dose Somatropin vs Label Dose Somatropin; Test type: Superiority or Other; p = 0.388, ANOVA — P-value for 12-Month Height SDS Change; Mean Difference (Net) = 0.16, 95% CI [-0.21 to 0.53] — Mean Difference = High Dose - Label Dose
Statistical Analysis 2: Comparison: High Dose Somatropin vs Label Dose Somatropin; Test type: Superiority or Other; p = 0.061, ANOVA — P-value for 24-Month Height SDS Change; Mean Difference (Net) = 0.49, 95% CI [-0.02 to 0.99] — Mean Difference = High Dose - Label Dose

3. Secondary Outcome: Height Velocity Standard Deviation Score (SDS) at 24 Month Endpoint
Description: as for outcome 1
Time Frame: 24 Months
Population: All enrolled participants with at least one post-baseline height velocity measurement, using the last observation available prior to the 24-month visit if the 24-month height velocity was not available.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | High Dose Somatropin | Label Dose Somatropin
Number analyzed (Participants) | 13 | 11
standard deviation score | 2.58 (1.86) | 1.45 (1.06)
Statistical Analysis 1: Comparison: High Dose Somatropin vs Label Dose Somatropin; Test type: Superiority or Other; p = 0.088, ANOVA; Mean Difference (Net) = 1.13, 95% CI [-0.18 to 2.44] — Mean Difference = High Dose - Label Dose

ADVERSE EVENTS:
Arm/Group | High Dose Somatropin | Label Dose Somatropin
Serious Adverse Events (participants affected / at risk) | 1 | 0
Other Adverse Events (participants affected / at risk) | 13 | 5
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | High Dose Somatropin | Label Dose Somatropin
Vertebral injury (Injury, poisoning and procedural complications) | 1/14 (1) | 0/13 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | High Dose Somatropin | Label Dose Somatropin
Anaemia (Blood and lymphatic system disorders) | 1/14 (1) | 0/13 (0)
Retinoschisis (Eye disorders) | 0/14 (0) | 1/13 (1)
Chest pain (General disorders) | 1/14 (1) | 0/13 (0)
Pyrexia (General disorders) | 2/14 (2) | 2/13 (2)
Ear infection (Infections and infestations) | 1/14 (2) | 0/13 (0)
Genital infection (Infections and infestations) | 0/14 (0) | 1/13 (1)
Impetigo (Infections and infestations) | 1/14 (1) | 0/13 (0)
Influenza (Infections and infestations) | 2/14 (3) | 0/13 (0)
Pharyngitis (Infections and infestations) | 1/14 (6) | 1/13 (1)
Rhinitis (Infections and infestations) | 1/14 (1) | 0/13 (0)
Varicella (Infections and infestations) | 1/14 (1) | 1/13 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1/14 (1) | 0/13 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 1/14 (1) | 0/13 (0)
Insulin resistance (Metabolism and nutrition disorders) | 2/14 (2) | 0/13 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 0/13 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 0/13 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 2/14 (2) | 0/13 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/14 (2) | 1/13 (1)
Disturbance in attention (Nervous system disorders) | 1/14 (1) | 0/13 (0)
Headache (Nervous system disorders) | 3/14 (10) | 0/13 (0)
Syncope (Nervous system disorders) | 1/14 (1) | 0/13 (0)
Epididymal cyst (Reproductive system and breast disorders) | 1/14 (1) | 0/13 (0)
Gynaecomastia (Reproductive system and breast disorders) | 3/14 (3) | 1/13 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/14 (0) | 1/13 (1)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1/14 (1) | 0/13 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1/14 (2) | 0/13 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days